CLINICAL TRIAL: NCT02490982
Title: Teriflunomide Observational Effectiveness Study
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Montreal Neurological Institute and Hospital (Other)
Responsible Party: Principal Investigator, Pierre Duquette, MD, Centre hospitalier de l'Université de Montréal (CHUM)
Other Study IDs: CE15.016
Record Dates: First submitted 2015-06-26; First posted 2015-07-07 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — teriflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Teriflunomide: Patient-reported outcomes and clinical assessment
  Interventions: Drug: Teriflunomide

INTERVENTIONS:
Drug: Teriflunomide — The prescription of Teriflunomide administered orally as a 14mg daily compound to RRMS patients.
  Other Names: Aubagio

SUMMARY:
The main goal of this investigator-initiated study is to evaluate the effectiveness and efficacy of Teriflunomide in a population of Relapsing Remitting Multiple Sclerosis (RRMS) patients treated in regular practice, over a period of at least two years, in the regular setting of a Multiple Sclerosis Clinic.

DETAILED DESCRIPTION:
Consenting adult RRMS patients, meeting all inclusion criteria and who have been prescribed Teriflunomide by their treating physician will be asked to complete questionnaires on quality of life (QoL), fatigue, and employment.

The study will include 300 participants from three Multiple Sclerosis (MS) Clinics. Disease and magnetic resonance imaging (MRI) activity, blood tests (aspartate aminotransferase (AST), alanine aminotransferase (ALT), complete blood count (CBC)), drug compliance, side effects, toxicity, will be monitored.

MS patients never treated with a disease modifying drug (DMD) and MS patients previously exposed to another DMD will be included. Some would have been on a single medication, while others would have been treated with two or more medications.

The results of the study will provide the patient-perceived global impacts of Teriflunomide on the patient's overall quality of life.

These results will also guide the physician in giving a treatment that will be adapted to the patient's major concerns.

ELIGIBILITY:
Inclusion Criteria:

* Consenting Relapsing Remitting Multiple Sclerosis adults with an Expanded Disability Status Scale (EDSS) score ≤ 5.0 who have been prescribed Teriflunomide and who agree to follow study procedures.

Exclusion Criteria:

* Primary progressive or secondary progressive Multiple Sclerosis without relapses; other diseases that may confound evaluation of outcomes; other exclusion as per product monograph; and women contemplating pregnancy or actually pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Relapsing Remitting Multiple Sclerosis patients followed at three MS Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcome (PRO) scores | one year
  Change on patient-reported outcome measures, from baseline score and at each visit.

SECONDARY OUTCOMES:
Disease activity - Composite measure | one year
  Change in the annualized relapse-rate and the Expanded Disability Status Scale (EDSS) over the two year period.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Duquette, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Connor P, Wolinsky JS, Confavreux C, Comi G, Kappos L, Olsson TP, Benzerdjeb H, Truffinet P, Wang L, Miller A, Freedman MS; TEMSO Trial Group. Randomized trial of oral teriflunomide for relapsing multiple sclerosis. N Engl J Med. 2011 Oct 6;365(14):1293-303. doi: 10.1056/NEJMoa1014656. PMID 21991951
- [Background] Rush AJ. The role of efficacy and effectiveness trials. World Psychiatry. 2009 Feb;8(1):34-5. doi: 10.1002/j.2051-5545.2009.tb00206.x. No abstract available. PMID 19293957
- [Background] Deshpande PR, Rajan S, Sudeepthi BL, Abdul Nazir CP. Patient-reported outcomes: A new era in clinical research. Perspect Clin Res. 2011 Oct;2(4):137-44. doi: 10.4103/2229-3485.86879. PMID 22145124
- [Background] Basch E. Toward patient-centered drug development in oncology. N Engl J Med. 2013 Aug 1;369(5):397-400. doi: 10.1056/NEJMp1114649. Epub 2013 Jul 3. No abstract available. PMID 23822654
- [Background] Nortvedt MW, Riise T. The use of quality of life measures in multiple sclerosis research. Mult Scler. 2003 Feb;9(1):63-72. doi: 10.1191/1352458503ms871oa. PMID 12617271
- [Background] Teriflunomide (Aubagio) (14 mg Film-coated Tablet): Teriflunomide is Indicated as Monotherapy for the Treatment of Patients with Relapsing-Remitting Multiple Sclerosis to Reduce the Frequency of Clinical Exacerbations and to Delay the Accumulation of Physical Disability [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2014 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK253634/ PMID 25411660